CLINICAL TRIAL: NCT00714389
Title: Uroflow Measurements in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Gunhilde Buchsbaum, MD, University of Rochester
Other Study IDs: 22847
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Results first posted 2010-01-29 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Urogynecology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study to determine normal values for certain urinary measurements in order to better understand voiding dysfunction in women.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers/employees
* Normal voiding function.
* Willing to participate.

Exclusion Criteria:

* Subjects currently receiving treatment for any lower urinary tract condition or having any voiding difficulty.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Urogynecology clinic
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gunhilde Buchsbaum, MD, Principal Investigator — University of Rochester
Locations (1):
- Urogynecology and Reconstructive Pelvic Surgery Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Urogynecology and OBGYN clinic March 2008
Groups:
- Spontaneous Uroflow Measurements: Spontaneous voids of volunteers working in the care facility will recorded by uroflowmetry.
Period: Overall Study
Arm/Group | Spontaneous Uroflow Measurements
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Spontaneous Uroflow Measurements: Spontaneous voids of subjects were recorded using uroflowmetry.
Arm/Group | Spontaneous Uroflow Measurements
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 50 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Voided Volume
Description: Volume of spontaneous void
Time Frame: March 2008
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Spontaneous Uroflow Measurements
Number analyzed (Participants) | 12
mL | 306 (148)

2. Primary Outcome: Maximal Flow Rate
Description: Maximal uroflow of spontaneous subject voids
Time Frame: March 2008
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | Spontaneous Uroflow Measurements
Number analyzed (Participants) | 12
mL/sec | 49 (16)

ADVERSE EVENTS:
Arm/Group | Spontaneous Uroflow Measurements
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Limited number of participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No